CLINICAL TRIAL: NCT05586815
Title: Efficacy of Colistin Monotherapy Versus Colistin Plus Minocycline for Therapy of Carbapenem-Resistant Acinetobacter Baumannii Infection
Brief Title: Efficacy of Colistin Monotherapy Versus Colistin Plus Minocycline for Carbapenem-Resistant A. Baumannii Infection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SI-CEU-03-2022
Record Dates: First submitted 2022-10-17; First posted 2022-10-19 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Acinetobacter Infections
Keywords: colistin; minocycline; carbapenem-resistant Acinetobacter baumannii
MeSH Terms: conditions — Acinetobacter Infections; cyclopia sequence | interventions — Colistin; colistinmethanesulfonic acid; Minocycline

STUDY DESIGN:
Intervention Model Description: A Phase 4 Randomized, Double blind, Placebo Controlled
Who Masked: Participant, Investigator
Masking Description: Double blind, Placebo Controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colistin plus Placebo (Active Comparator): Colistin alone, 150 mg every 8 hours intravenously or according to renal function, plus Placebo
  Interventions: Drug: Colistin; Drug: Placebo
- Colistin plus Minocycline (Experimental): Colistin, 150 mg every 8 hours intravenously or according to renal function, plus Minocycline, 200 mg every 12 hours orally
  Interventions: Drug: Colistin; Drug: Minocycline

INTERVENTIONS:
Drug: Colistin — 150 mg every 8 hours intravenously for at least 7 and up to a maximum of 28 days
  Other Names: Sodium colistimethate
Drug: Minocycline — 200 mg every 12 hours orally for at least 7 and up to a maximum of 28 days
  Other Names: Mino
  Arms: Colistin plus Minocycline
Drug: Placebo — Capsule without active compound
  Arms: Colistin plus Placebo

SUMMARY:
Acinetobacter baumannii causes severe infections (pneumonia, bacteremia, organ space) with high lethality in hospitalised critically ill patients. It can acquire resistance to all classes of antibiotics (multidrug resistance, MDR) except an 'old' drug, colistin, which may be the only therapeutic option. The addition of minocycline to colistin has been shown to be synergistic in vitro, and may be promising in vivo, but this combination has not been limited to case report or case series in comparison with colistin alone.

DETAILED DESCRIPTION:
The purpose of this double-blind, randomized, parallel, placebo-controlled clinical trial is to assess whether the association of colistin and minocycline reduces significantly the mortality of patients with severe MDR A. baumannii infections compared with colistin alone.

The trial will enroll 94 patients from internal medicine ward and intensive care units (ICU) of an university care hospitals where MDR A. baumannii infection is endemic with epidemic phases. Patients will be randomly allocated to either colistin plus placebo (control arm) or colistin plus minocycline (experimental arm).

Primary end point is overall mortality, defined as death occurring within 28 days from randomisation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and microbiological evidence of a severe infection due to multi-drug resistant A. baumannii during hospitalization
* Susceptibility of the A. baumannii isolate to colistin (MIC < or =2 mg/l).

Exclusion Criteria:

* Treatment with one of the study drugs prior to the diagnosis of A. baumannii infection more than 48 hours
* Severe liver dysfunction
* History of prior hypersensitivity to the study drugs
* Pregnancy and lactation

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | 28 days
  The study primary outcome is patient overall mortality, defined as death occurring during hospitalisation or within 28 days from randomization.

SECONDARY OUTCOMES:
Microbiological eradication | 28 days
  Microbiological eradication is defined as the disappearance of A. baumannii in cultures from blood, bronchial aspirate, urines and drainage fluids.
Incidence of Renal toxicity (safety) | 28 days
  Renal toxicity is defined as decrease of creatinine clearance below 50 ml/min or >50% reduction in the creatinine clearance relative to the baseline.
Incidence of Hepatic toxicity (safety) | 28 days
  Hepatic toxicity is defined as increase of direct bilirubin above 3 mg/dl.

CONTACTS AND LOCATIONS:
Overall Officials: Adhiratha Boonyasiri, MD, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koomanachai P, Tiengrim S, Kiratisin P, Thamlikitkul V. Efficacy and safety of colistin (colistimethate sodium) for therapy of infections caused by multidrug-resistant Pseudomonas aeruginosa and Acinetobacter baumannii in Siriraj Hospital, Bangkok, Thailand. Int J Infect Dis. 2007 Sep;11(5):402-6. doi: 10.1016/j.ijid.2006.09.011. Epub 2007 Feb 8. PMID 17291803
- [Background] Thamlikitkul V, Tiengrim S, Seenama C. Comparative in vitro activity of minocycline and selected antibiotics against carbapenem-resistant Acinetobacter baumannii from Thailand. Int J Antimicrob Agents. 2016 Jan;47(1):101-2. doi: 10.1016/j.ijantimicag.2015.11.006. Epub 2015 Dec 11. No abstract available. PMID 26725031